CLINICAL TRIAL: NCT04179253
Title: Hysteroscopic Evaluation of Uterine Cavity in Women With Unexplained Infertility
Brief Title: Detection of the Uterine Abnormalities Missed in an Ultrasound Scan and/or Hysterosalpingography Using Hysteroscopy, in Females Presenting With Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Associate Professor in Obstetrics and Gynecology Department, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Beni-Suef 19
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: One hundred women with unexplained infertility recruited for office micro hysteroscopic session
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unexplained infertility (Other): The patient was placed in the dorsal lithotomy position. Normal saline was used for uterine distension connected to the inflow channel on the sheath with intravenous tubing. The tip of the hysteroscope was positioned in the vaginal introitus, the labia being slightly separated with fingers. The vagina was distended with saline.
  The uterine cavity was systematically explored by rotating the fore-oblique scope in order to identify any anomaly in the uterine walls and/or the right and left tubal ostia. At this stage it was crucially important to avoid lateral movements as much as possible to reduce patient discomfort to a minimum. After that, the scope was removed Finally the evaluation and the data that had been found were written in details by the surgeon. Operative intervention was done if needed. Any complication in the form of pain, bleeding, vasovagal attack and perforation, were registered in the patient sheet.
  Interventions: Diagnostic Test: office micro hysteroscopy

INTERVENTIONS:
Diagnostic Test: office micro hysteroscopy — One hundred women with unexplained infertility recruited for office micro hysteroscopic sessions. A rigid fiberoptic 2-mm, 0 and 30 degrees angled hysteroscopy along with an operative channel for grasping forceps or scissors were used for both diagnostic and operative indications. The findings, complications, and patient tolerance were recorded.

SUMMARY:
Hysteroscopy is still considered the gold standard procedure for uterine cavity exploration. Therefore, many specialists have used hysteroscopy as their first-line of routine exam for infertility patients regardless of guidelines. Thus, scheduling the office micro hysteroscopy as one of the routine steps in the fertility workup program has become mandatory before the final diagnosis of unexplained infertility.

DETAILED DESCRIPTION:
Although hysteroscopy is generally accepted as the gold standard in diagnosis and treatment of uterine cavity pathology, many gynecologist are reluctant to perform hysteroscopy as an initial test without a high degree of suspicion for pathology due to the need for anesthesia in an operating room setting. The basic infertility work-up has included a HSG to evaluate the uterine cavity and tubal patency. However, HSG does not allow for simultaneous correction of uterine pathology. Moreover HSG may miss 35% of uterine abnormalities. Hysterolaparoscopy (Pan Endoscopic) approach is better than HSG and should be encouraged as first and final procedure in selected infertile women.

Sonohysterography (SHG) has been proposed as a better diagnostic test of the uterine cavity. However, it also suffers from a sensitivity and specificity inferior to that of hysteroscopy in most studies.

ELIGIBILITY:
Inclusion Criteria:

* Normal HSG
* Normal Ultrasound
* Normal Hormonal Profile
* Normal Semen

Exclusion Criteria:

* Abnormal findings in different investigations of infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-14 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Abnormal hysteroscopic findings | one year
  Description of different hysteroscopic abnormalities using micro-office hysteroscope

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper NA, Smith P, Khan KS, Clark TJ. A systematic review of the effect of the distension medium on pain during outpatient hysteroscopy. Fertil Steril. 2011 Jan;95(1):264-71. doi: 10.1016/j.fertnstert.2010.04.080. Epub 2010 Jun 23. PMID 20576262
- [Background] Molinas CR, Campo R. Office hysteroscopy and adenomyosis. Best Pract Res Clin Obstet Gynaecol. 2006 Aug;20(4):557-67. doi: 10.1016/j.bpobgyn.2006.01.019. Epub 2006 Mar 22. PMID 16554185
- [Background] Vaid K, Mehra S, Verma M, Jain S, Sharma A, Bhaskaran S. Pan endoscopic approach "hysterolaparoscopy" as an initial procedure in selected infertile women. J Clin Diagn Res. 2014 Feb;8(2):95-8. doi: 10.7860/JCDR/2014/7271.4018. Epub 2014 Feb 3. PMID 24701493
- [Background] Kowalczyk D, Guzikowski W, Wiecek J, Sioma-Markowska U. Clinical value of real time 3D sonohysterography and 2D sonohysterography in comparison to hysteroscopy with subsequent histopathological examination in perimenopausal women with abnormal uterine bleeding. Neuro Endocrinol Lett. 2012;33(2):212-6. PMID 22592204